CLINICAL TRIAL: NCT02991131
Title: DART: "Sivextro® in Acute Bacterial Skin anD Skin Structure Infection (ABSSSI) in Hospitalized Patients. A Global ObseRvational STudy."
Brief Title: Sivextro in Acute Bacterial Skin and Skin Structure Infection (ABSSSI) in Hospitalized Patients. A Global Observational Study
Acronym: DART
Status: Terminated | Type: Observational
Why Stopped: Company decision
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18299; SX1601 (Other: Company Internal)
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Skin Disease, Infectious
Keywords: Acute bacterial skin infection; Acute Bacterial Skin and Skin Structure Infection (ABSSSI); Abscess; Cellulitis; Erysipelas; Wound infection; Methicillin resistant Staphylococcus aureus (MRSA)
MeSH Terms: conditions — Skin Diseases, Infectious; Abscess; Cellulitis; Erysipelas; Wound Infection | interventions — tedizolid; tedizolid phosphate; Linezolid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tedizolid: Hospitalized ABSSSI patients treated with tedizolid
  Interventions: Drug: Tedizolid (Sivextro, BAY1192631)
- Linezolid: Hospitalized ABSSSI patients treated with linezolid
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Tedizolid (Sivextro, BAY1192631) — Antibiotic
  Groups: Tedizolid
Drug: Linezolid — Antibiotic
  Groups: Linezolid

SUMMARY:
This open-label, prospective, multi-center, non-interventional, observational, parallel cohort study intended to provide real life data on the treatment duration, effectiveness and safety of tedizolid and linezolid when treating ABSSSI hospitalized patients in a real practice setting.

DETAILED DESCRIPTION:
The primary objective of this study was to assess the treatment duration in the real life in 2 cohorts consisting of patients treated by 200 mg once daily IV/PO tedizolid or treated by 600 mg twice daily IV/PO (intravenous/per oral) linezolid.

ELIGIBILITY:
Inclusion Criteria:

* Adult female and male in-patients with clinical diagnosis compatible with ABSSSI (cellulitis/erysipelas, major skin abscess or wound infections) with a clinical suspicion of infection by Gram positive bacteria (with or without laboratory confirmation).
* Patients for whom the decision to initiate treatment with tedizolid phosphate or linezolid was made as per physician's routine treatment practice.
* Signed informed consent.

Exclusion Criteria:

* Patients participating in an investigational program with interventions outside of routine clinical practice.
* Patients who have been enrolled in this study before.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2016-12-17 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Number of treatment days | Up to 1 month
  Duration of treatment is defined as the time interval from date of first administration of tedizolid or linezolid to the date of permanent discontinuation of tedizolid or linezolid, respectively.
  The treatment is according to the recommendations written in the local product information.

SECONDARY OUTCOMES:
Number of participants with adverse events or safety-relevant changes in laboratory parameters | Up to 1 month

OTHER OUTCOMES:
Number of participants with investigator-assessed clinical response | Up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Multiple Locations, Mexico
- Multiple Locations, Russia
- Multiple Locations, Singapore